CLINICAL TRIAL: NCT06188663
Title: SalT Supplementation in Older Adults With Orthostatic Intolerance Disorders (STOOD): a Phase IIa Randomised Controlled Trial of Sodium Supplementation in Those Consuming Moderate Salt Intake.
Brief Title: SalT Supplementation in Older Adults With Orthostatic Intolerance Disorders
Acronym: STOOD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Galway (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Catriona Reddin, Research Fellow, Geriatric Medicine SpR, University of Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.A.3086
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Orthostatic Hypotension
Keywords: Orthostatic Hypotension; Sodium; Diet
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Masking Description: This study is open-label. Blinding of participants is not possible for practical reasons. However, there is blinded assessment of change in formula derived 24-hour urinary sodium, cardiovascular biomarkers and mean 24-hour ambulatory blood pressure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt supplementation (Active Comparator): Salt supplementation in the form of 1.25g sodium chloride capsules at a dose of 5g/day in two divided doses
  Interventions: Dietary Supplement: Salt supplementation (encapsulated sodium chloride)
- Usual salt intake (no change in intake) (No Intervention): Usual salt intake (no change in intake)

INTERVENTIONS:
Dietary Supplement: Salt supplementation (encapsulated sodium chloride) — A high salt intake range will be achieved through unchanged dietary intake and supplementary salt in the form of 1.25g sodium chloride capsules at a dose of 5g/day in two divided doses
  Arms: Salt supplementation

SUMMARY:
Background

Orthostatic hypotension (OH) is a common cause of falls, and key source of morbidity and mortality due to injury (e.g. hip fracture). Current guidelines recommend increasing salt intake in patients with symptomatic orthostatic hypotension. However, the evidence underpinning this recommendation is poor, based primarily on small trials with very short-term follow-up (< 6 weeks).

Clinical Equipoise (Overall)

High salt intake might improve quality of life and reduce the risk of falls, but might also increase the risk of cardiovascular disease, in patients with OH.

Specific Objective of Current Application (Aim)

To determine feasibility (recruitment, retention and adherence) of conducting a randomized controlled trial evaluating high salt intake in older adults with symptomatic orthostatic hypotension.

To determine preliminary estimates of the effect of high salt intake on disease-specific quality of life, orthostatic blood pressure (BP) parameters, and cardiac blood biomarkers.

Design: Phase IIa, parallel, double-blind, randomised controlled, single centre clinical trial of 12 month follow-up duration.

Population: Older adults (≥65 years of age) with an objective diagnosis of symptomatic orthostatic hypotension

Intervention: The intervention will be 5g/day of salt supplementation in the form of encapsulated sodium chloride.

Outcome measures: Primary outcome (Feasibility) recruitment and retention rates, adherence with intervention and study protocol, completeness of follow-up. Secondary Outcome (Efficacy): i) clinical: change in Orthostatic Hypotension Questionnaire score, modification/addition of OH pharmacotherapy, and falls events, ii) physiological measures of orthostasis: change in difference between supine and nadir systolic BP, standing BP at 1 minute, 24 hour mean BP measured by 24 hour ambulatory BP monitor, iii) cardiovascular biomarkers.

Clinical Importance:

A recommendation for long-term increases in salt intake may have adverse cardiovascular consequences, which necessitates the identification of the optimal range of salt intake associated with greatest reduction in falls risk and lowest cardiovascular risk. Our study will provide preliminary evidence of treatment effect and assess feasibility, to inform a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 65 years of age
* Documented history of orthostatic hypotension, defined by decrease in systolic blood pressure (SBP) of ≥20 mmHg or a decrease in diastolic blood pressure (DBP) of ≥10 mmHg within three minutes of standing when compared with blood pressure from the supine position, or at head-up tilt testing.
* A documented history of symptoms consistent with orthostatic hypotension including one of the following: light-headedness, dizziness, feeling faint, feeling like they may black out
* Baseline salt intake expected to be in the moderate range (5-10g/day) based on screening questions
* Willingness to supplement sodium intake
* Ability to provide written informed consent

Exclusion Criteria:

* Severe supine hypertension (Systolic blood pressure≥180mmHg or diastolic blood pressure >110mmHg) measured as average of three office readings
* A diagnosis of Heart Failure (New York Heart Association (NYHA) Class III or IV symptoms or known left ventricular ejection fraction 30%, if more than one echo eligibility is defined by most recent echo)
* CKD (eGFR <30ml/min/1.73m2) based on eGFR measured within the last 6 months
* Participants taking loop diuretics
* Serum sodium <125mmol at last measurement
* Acute intercurrent illness
* Prescribed high-salt diet (for clinical indication other than for OH) or low-salt diet for evidence based clinical indication
* Participant unlikely to comply with study procedures or follow-up visits due to severe comorbid illness or other factor (e.g. inability to travel for follow-up visits) in opinion of research team
* Inability to provide informed consent in the opinion of the investigator (for example due to severe cognitive impairment)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment to target (primary feasibility outcome) | 15 months
  Recruitment of 48 participants
Change in orthostatic hypotension questionnaire score (primary efficacy outcome) | 6 months
  Change in symptoms and quality of life measured using disease specific questionnaire; Orthostatic Hypotension Questionnaire (OHQ) from baseline to final follow-up. All questionnaire items are scored 0 through 10 (higher scores = worse).

SECONDARY OUTCOMES:
Change in individual components of OHQ from baseline to final follow-up | 6 months
  Change in individual components of OHQ from baseline to final follow-up. All questionnaire items are scored 0 through 10 (higher scores = worse).
Rates of modification/addition of OH pharmacotherapy | 6 months
  Rates of modification/addition of OH pharmacotherapy
Rates of modification/addition of anti-hypertensive therapy | 6 months
  Rates of modification/addition of anti-hypertensive therapy
Falls events | 6 months
  Number of falls events
Change in difference between supine and nadir blood pressure from baseline to final in-person follow-up | 6 months
  Change in difference between supine and nadir blood pressure from baseline to final in-person follow-up
Change in standing BP at one minute and three minutes | 6 months
  Change in standing BP at one minute and three minutes measured at active stand
Change in mean BP measured by 24 hour ambulatory BP monitor | 6 months
  Change in mean BP measured by 24 hour ambulatory BP monitor
Change in cardiovascular biomarkers; proBNP and troponin | 6 months
  Change in cardiovascular biomarkers; proBNP and troponin
Change in formula derived 24 hour urinary sodium from baseline to final in-person follow-up visit. | 6 months
  Change in formula derived 24 hour urinary sodium
Change in renin-aldosterone ratio from baseline to final in-person follow-up visit. | 6 months
  Change in renin-aldosterone ratio from baseline to final in-person follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Martin O'Donnell, Principal Investigator — University of Galway; Catriona Reddin, Principal Investigator — University of Galway; Andrew Smyth, Principal Investigator — University of Galway
Locations (1):
- Clinical Research Facility Galway/Galway University Hospital, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No